CLINICAL TRIAL: NCT06236022
Title: The Effects of Sirolimus in Patients With Dilated Cardiomyopathy Infected With Kaposi Sarcoma-associated Virus
Acronym: SDCMK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Wuhan Central Hospital (Other); Wuhan Fourth Hospital (Unknown); Wuhan University (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Prof., Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJH-SDCMK
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Dilated Cardiomyopathy; Kaposi's Sarcoma-Associated Herpesvirus Infection
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): patients with dilated cardiomyopathy infected with Kaposi sarcoma-associated virus to receive standard DCM therapy
- Sirolimus (Experimental): patients with dilated cardiomyopathy infected with Kaposi sarcoma-associated virus to receive sirolimus (at a dose of 2 mg once daily) in addition to standard DCM therapy
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — at a dose of 2 mg once daily
  Arms: Sirolimus

SUMMARY:
Evaluating the efficacy of sirolimus (compared to standard therapy alone) in the treatment of dilated cardiomyopathy infected with Kaposi Sarcoma-associated virus -- a multicenter randomized controlled study.

DETAILED DESCRIPTION:
Dilated cardiomyopathy (DCM), defined as left ventricular or biventricular dilation and systolic dysfunction in the absence of either pressure or volume overload or coronary artery disease sufficient to explain the dysfunction, is associated with poor cardiovascular outcome and poor prognosis. Inflammation, activated by viral persistence, was considered as a key trigger factor of cardiac remodeling and thereby the development of DCM. As a risk factor for DCM, Kaposi's sarcoma-associated herpes virus (KSHV) inhibits the type I IFN signaling pathway and thereby aggravates known cardiotropic viruses-induced cardiac dysfunction and inflammatory infiltration. Activated mTOR signaling pathway is a typical feature of KSHV-infected cells, which is the most effective therapeutic target of diseases caused by KSHV infection. Sirolimus, a mTOR inhibitor, is a drug that can effectively treat the KSHV-infected diseases and suppresses the replication of KSHV.Therefore, multicenter large randomized controlled trials are needed to verify the efficacy of sirolimus on patients with DCM infected with KSHV.

This study aimed to evaluate the effiects of sirolimus on the clinical outcomes of patients with DCM infected with KSHV and provide theoretical evidence for the clinical application of sirolimus in these patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age;
* Diagnosed as dilated cardiomyopathy. Specifically, (i) left ventricular ejection fraction <45% (>2 SD) and/or fractional shortening <25% (>2 SD), as ascertained by echocardiography, radionuclide scanning, or cardiac magnetic resonance imaging; (ii) left ventricular end-diastolic diameter >117% of the predicted value corrected for age and body surface area (Henry's formula), which corresponds to 2 SD of the predicted normal limit +5%; and (iii) In the absence of severe coronary artery disease or valvular disease.
* KSHV DNA seropositivity;
* Patients are voluntary and signed informed consent.

Exclusion Criteria:

* Allergic to rapamycin or its derivatives；
* The proportion of neutrophils less than 0.5*10^9/L or platelet less than 2.5*10^10/L;
* Pregnant women or plan to;
* Participate in any drug clinical trials within 3 months;
* Serious neurological disease (Alzheimer's disease, Parkinson syndrome, progressive lower limbs or deaf patients);
* Previous history of cancer or tumor, or pathological examination confirmed precancerous lesions;
* Patients were not optimally managed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac mortality | up to 36 months
  Death from cardiovascular disease which includes coronary artery diseases, stroke, heart failure, hypertensive heart disease, rheumatic heart disease, cardiomyopathy, heart arrhythmia, congenital heart disease, valvular heart disease and carditis
Rate of heart transplantation | up to 36 months
  The rate of heart trans plantation on patients with DCM when other medical or surgical treatments have failed

SECONDARY OUTCOMES:
Readmission rate for cardiovascular diseases | up to 36 months
  The readmission rate for cardiovascular diseases
Recurrence rate of heart failure | up to 36 months
  The recurrence rate of heart failure
All-cause mortality | up to 36 months
  Death from all diseases
KCCQ score | up to 36 months
  The score of patients measured with the Kansas City Cardiomyopathy Questionnaire (KCCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China